CLINICAL TRIAL: NCT05286775
Title: The Functional Treatment of Disabling Pain in Knee Osteoarthritis in a Rehabilitation Program for the Brazilian Unified Health System
Brief Title: Knee Osteoarthritis Disabling Pain Program for the Brazilian Unified Health System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Imamura (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor-Investigator, Marta Imamura, MD PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08756819.8.0000.0068
Record Dates: First submitted 2022-02-11; First posted 2022-03-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Physical and Rehabilitation Medicine; Knee Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical treatment and Knee educational program (Experimental): Medical knee treatment combined with knee educational educational program
  Interventions: Other: Clinical treatment and Knee educational program
- Knee educational program (Active Comparator): Knee educational program
  Interventions: Other: Clinical treatment and Knee educational program; Other: Knee educational program

INTERVENTIONS:
Other: Clinical treatment and Knee educational program — Three weekly medical interventions, according to the patient's need as observed at baseline.
  1. 3ml paraspinal infusion of 1% Lidocaine (segmental spinal level);
  2. 5,000 impulses of Radial Shockwave Therapy (pneumatic generator, 0.16mJ/mm² of energy and 20Hz of frequency) at the most painful spot of the knees;
  3. *6,000 pulses of Focused Shockwave Therapy (electromagnetic generator) at four sites of the painful knee.
     For those with knee pain of 7 or above in Visual Analogue Scale after the treatments above, the interventions below will be delivered in the order they appear:
  4. Ultrasound guided genicular nerve block: infusion of up to 10ml 0.50% Levobupivacaine without vasoconstrictor;
  5. Hydrodissection of superficial and deep plane nerves: infusion of 10ml 5% dextrose diluted in water (D5W);
  6. Intra-articular Infusion of Hyaluronic Acid: ultrasound guided infusion of 2.5ml of sodium hyaluronate at the knee joint.
     * Four weekly applications.
Other: Knee educational program — Three weekly 60-minute educational program sessions with the following services:
  Stretching and strengthening exercises for specific muscle groups (hip flexors, extensors, and abductors; knee flexors and extensors; plantar flexors; and abdominal muscles), using one's own body and gravity resistance. Patients will be encouraged to practice them at home at least twice a week after the end of the sessions.
  Nutritional guidance: Instructions on the importance of adequate weight management, healthy food consumption, and the adequate intake of nutrients.
  Physical activities: Counseling on home-based physical activities, according to their physical capacities, to protect knee joints.
  General health: psychology counseling, encouraging participants to apply strategies and self help conduct to improve their general health; Occupational Therapy: Activities of Daily Living strategies to protect knee joints; Nursing: Counseling on strategies for improving healthy sleeping habits.
  Arms: Knee educational program

SUMMARY:
This is a Randomized Clinical Trial to compare two interventions for reducing knee pain and improving knee function of patients with knee osteoarthritis.

Sixty participants will be randomly allocated to one of the intervention groups, either a knee educational program or a combination of knee educational program and medical interventions.

Participants will be assessed primarily on function and pain, as well as other secondary outcomes at baseline, at the end of the interventions, and three months after the end of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee osteoarthritis;
* Moderate to severe knee pain (VAS >= 4);
* Knee pain for at least 3 months prior to inclusion;
* Willing to sign the Informed Consent Form.

Exclusion Criteria:

* Untreated severe psychological or psychiatric diseases without treatment;
* Presence of fibromyalgia;
* Presence of systemic inflammatory rheumatic diseases;
* Presence of neoplasia;
* Presence of relevant pain in other joints, according to medical evaluation;
* Presence of intolerance or allergy to Lidocaine or local anaesthetics;
* Concomitant use of anticoagulant drug.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Knee function | Baseline and up to six months from baseline.
  Change of knee function from baseline measured with Knee Injury and Osteoarthritis Outcome Score (KOOS)

SECONDARY OUTCOMES:
Knee function | Baseline and up to three months from baseline.
  Change of knee function from baseline measured with Knee Injury and Osteoarthritis Outcome Score (KOOS)
Knee pain as assessed by Visual Analogue Scale (VAS) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of knee pain from baseline measured with Visual Analogue Scale (VAS), a 0 - 10 rating scale in which 0 means no pain and 10 means the worst pain possible.
Quality of Life Assessment as assessed by the 36-Item Short-Form Health Survey (SF-36) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of Quality of Life from baseline measured with the 36-Item Short-Form Health Survey (SF-36)
Physical activity level | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of classification of physical activity level according to a physical activity level scale
Pain pressure threshold | Baseline, end of treatment, and three months from end of treatment.
  Change of pain pressure threshold measured bilaterally with an algometer, at vastus medialis, adductor longus, rectus femoris, vastus lateralis, tibialis anterior, peroneus longus, iliacus, sartorius, gracilis, quadratus lumborum, popliteus, and ligaments located over the supraspinous ligaments between L1-L2, L2-L3, L3-L4, L4-L5, L5-S1 and sacral (S) areas S1-S2.
Pain modulation | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of conditioned pain modulation test of hands in cold water
Bio-mechanical assessment (Steps) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of bio-mechanic variables, assessment with a wearable three axial accelerometer. The patients will wear an accelerometer (Actigraph) for one week before all evaluation time points. Daily data on number of steps will be collected.
Bio-mechanical assessment (Energy Expenditure) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of bio-mechanic variables, assessment with a wearable three axial accelerometer. The patients will wear an accelerometer (Actigraph) for one week before all evaluation time points. Daily data on energy expenditure (kcal) will be collected.
Bio-mechanical assessment (Physical activity intensity) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of bio-mechanic variables, assessment with a wearable three axial accelerometer. The patients will wear an accelerometer (Actigraph) for one week before all evaluation time points. Daily data on physical activity intensity will be collected.
Bio-mechanical assessment (Step velocity) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change of bio-mechanic variables, assessment with a wearable three axial accelerometer. The patients will wear an accelerometer (Actigraph) for one week before all evaluation time points. Daily data on step velocity (steps/second) will be collected.
Gait analysis (gait cycle) | Baseline and up to three months from baseline.
  Change of gait parameters measured by a three-dimensional gait analysis system in a gait analysis lab. Ten Infra-red cameras will detect gait parameters and a platform will detect the different pressures delivered by both lower limbs during gait. Bilateral gait cycle (seconds) will be collected, compared and analyzed.
Gait analysis (joint angles) | Baseline and up to three months from baseline.
  Change of gait parameters measured by a three-dimensional gait analysis system in a gait analysis lab. Ten Infra-red cameras will detect gait parameters and a platform will detect the different pressures delivered by both lower limbs during gait. Bilateral joint angles (degrees) will be collected and analyzed.
Muscle strength (Work) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change in muscle strength (knee flexion and extension) measured by an isokinetic dynamometry (Cybex), at 60º and 120º per second. The analyzed variables will be work (Joules - J).
Muscle strength (Power) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change in muscle strength (knee flexion and extension) measured by an isokinetic dynamometry (Cybex), at 60º and 120º per second. The analyzed variables will be Power (Watts - W).
Muscle strength (Peak torque) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change in muscle strength (knee flexion and extension) measured by an isokinetic dynamometry (Cybex), at 60º and 120º per second. The analyzed variables will be bilateral Peak tork (Newton meters - Nm).
Muscle strength (Agonist/Antagonist Balance) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change in muscle strength (knee flexion and extension) measured by an isokinetic dynamometry (Cybex), at 60º and 120º per second. The analyzed variables will be agonist/antagonist balance of knee flexion and extension (difference of strength between agonist/antagonist in %).
Functional mobility | Baseline, up to three months from baseline, and up to six months from baseline.
  Change in functional mobility measured with the Timed Up and Go test (TUG)
Cutaneous temperature | Baseline, up to three months from baseline, and up to six months from baseline.
  Change in cutaneous temperature of the knee with Infra-red thermography images.

OTHER OUTCOMES:
Nutritional status | Baseline
  Nutritional status scale
Body Mass Index | Baseline
  Body Mass Index (BMI): the ratio of weight divided by the squared height.
Cognitive status | Baseline
  Cognitive status measured with Montreal Cognitive Assessment Test (MoCA)
Electroencephalogram (EEG) | Baseline, up to three months from baseline, and up to six months from baseline.
  Change from baseline of neurophysiological parameters with an EEG system. The analyzed parameters will be absolute power (μV2) and relative power (power in a specific frequency range/total power from 1 to 40 Hz) for the frequency bands delta (1-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), and the sub-bands: low beta (13-20 Hz) and high beta (20-30 Hz), measured at the central, parietal, and frontal areas.
Magnetic Resonance Imaging (MRI) | Baseline
  Magnetic resonance imaging of the knees
Demography | Baseline
  Demographic characteristics of participants, such as age, sex, schooling, body mass index (BMI), concomitant medical drug use, and comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Medicina Física e Reabilitação (IMREA-FMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) may be shared in the future under suitable request and justification to principal investigator.